CLINICAL TRIAL: NCT00650897
Title: Escitalopram Treatment of Major Depression in Diabetes Mellitus: An Open Label
Brief Title: Efficacy Study of Escitalopram for Depression in Patients With Diabetes
Acronym: EFDID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Raz Gross, The Gertner Institute for Epidemiology and Health Policy Research Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4426-RG-CTIL
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Major Depression; Diabetes Mellitus
Keywords: Efficacy; Antidepressant; Escitalopram; Major Depression; Diabetes Mellitus; Self Care
MeSH Terms: conditions — Depressive Disorder, Major; Diabetes Mellitus | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients with Diabetes Mellitus and Major Depression
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10-20 mg once daily

SUMMARY:
Patients with diabetes and major depression treated with Escitalopram might experience significant improvement in depression and anxiety scores; functional ability; diabetes-related self-care; and pain symptoms

DETAILED DESCRIPTION:
Major depression is common in patients diabetes (point prevalence about 15-20%). It has been shown that patients with diabetic and major depression experience more severe diabetes symptoms, greater disability, more frequent medical complications, greater healthcare utilization costs, poorer glycemic control, and greater difficulties with diabetes self-care activities, compared with patients with diabetes without depression. Few specific features of Escitalopram, a selective serotonin reuptake inhibitor (SSRI), make it a promising medication for use in diabetes. These include a benign side effect profile; high tolerance in elderly patients; rapid action with efficacy often demonstrated in as little 1-2 weeks, which in turn could help improve compliance; its efficacy for treatment of generalized anxiety disorder, which may also be relatively common in patients with diabetes, and co-occurs frequently with depression. This study is designed to test the efficacy of Escitalopram for the treatment of major depression in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosis of Type-1 or Type-2 diabetes mellitus (excluding gestational diabetes) by a specialist at least 6 months prior to the study.
* Current diagnosis of major depression based on DSM-IV criteria .
* Hamilton Depression Rating Scale (HAMD) baseline score > 17
* Available for 14-weeks of treatment and all evaluations.
* Able to understand study rules and procedures and willing to sign written informed consent for study participation.

Exclusion Criteria:

* Competence: Not competent to understand and sign informed consent forms and/or to understand and answer the evaluations.
* Psychiatric exclusions: One or more of the following: Alcohol or substance abuse or dependence in past 6 months; psychotic symptoms or history of psychosis; bipolar disorder; organic brain syndrome; significant suicide risk; homicidal thoughts.
* Medical exclusions: Known intolerance or hypersensitivity to escitalopram or other SSRI; pregnancy; breastfeeding; women of childbearing potential not using adequate contraception; significant renal or hepatic dysfunction (such that demands medical workup and/or regular follow up); resting heart rate less than 40/minute (or 50/minute if symptomatic); uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg); any acute or unstable medical condition that might interfere with the safe conduct of the study.
* Concomitant medication(s) exclusion: Current use (within 2 weeks of enrollment) of one or more of the following: antidepressants; regular benzodiazepine; neuroleptics; anticonvulsants; reserpine; guanethidine; clonidine; methyldopa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-06 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 14 weeks

SECONDARY OUTCOMES:
Diabetes self-care | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raz Gross, MD; MPH, Principal Investigator — The Gertner Institute
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel